CLINICAL TRIAL: NCT04116385
Title: Evaluation of the Quantra System in a Surgical Oncological Population
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-025
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Blood Loss, Surgical
Keywords: Viscoelastic testing; Coagulation; Quantra; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Cancer surgery patients: Adult subjects (18 years or older) undergoing an oncologic surgical procedure.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: Quantra QPlus System

SUMMARY:
This study will monitor coagulation parameters during the perioperative course of cancer surgical procedures using the Quantra System with the QPlus Cartridge.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The Quantra QPlus Cartridge was developed to monitor hemostasis during major surgical procedures in adult patients. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed iin parallel yielding six parameters that depict the functional status of a patient's coagulation system.

The oncologic surgical population presents unique challenges to providers who must distinguish between a cancer patient's increased tendency toward both thrombosis and hemorrhage. This single site prospective observational study in oncologic patients will give an insight into the coagulation status of critically ill cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >= 18 years
* Subject is diagnosed with cancer and is scheduled for surgical resection
* Subject is willing to participate, and he/she or a Legally Authorized Representative (LAR) has signed a consent form
* Surgical procedure to be performed has an anticipated blood loss (>500mL) based on historical data

Exclusion Criteria:

* Subject is younger than 18 years
* Subject or a subject's LAR is unable to provide written informed consent
* Subject is undergoing an emergent procedure.
* Subject is pregnant, has active liver disease, or severe renal dysfunction (creatinine clearance (CrCL)<30 mL/min)
* Subject has an extremely low platelet count (<40,000/uL)
* Subject is currently enrolled in a distinct study that might confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the clinical team, may pose additional risks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult subjects undergoing an oncologic surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time results to TEG R results | Baseline, defined as after induction of anesthesia, before surgical incision
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Stiffness results to TEG MA results | Baseline, defined as after induction of anesthesia, before surgical incision
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Time results to TEG R results | During surgery
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Stiffness results to TEG MA results | During surgery
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Time results to TEG R results | Post-surgery, while patient is in the ICU/PACU, usually within 24 hours of surgery
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Stiffness results to TEG MA results | Post-surgery, while patient is in the ICU/PACU, usually within 24 hours of surgery
  Coagulation function assessed by Quantra and TEG 5000

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No